CLINICAL TRIAL: NCT04093843
Title: Accelerated rTMS as a Treatment for Post-stroke Depression in the Subacute Phase: an Open Label Pilot Study
Brief Title: TMS for Post Stroke Depression
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Amelia Adcock (Other)
Responsible Party: Sponsor-Investigator, Amelia Adcock, Associate professor, West Virginia University
Organization: West Virginia University (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 1804090922
Record Dates: First submitted 2019-07-16; First posted 2019-09-18 (Actual); Results first posted 2022-04-29 (Actual); Last update posted 2022-04-29 (Actual); Status verified 2022-04

CONDITIONS: Post-stroke Depression

STUDY DESIGN:
Intervention Model Description: Open label
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (1):
- TMS (Experimental): Open label single arm study to determine safety and effectiveness of TMS for post stroke depression
  Interventions: Device: TMS

INTERVENTIONS:
Device: TMS — NeuroStar TMS Therapy

SUMMARY:
The purpose of this study is to find alternative treatments for patient's suffering from depression after having a stroke.This study aims to show that accelerated rTMS is a safe, effective,and convenient treatment for patient's suffering from post-stroke depression in the acute to subacute phase. This will be an open label trial and thus all participants will receive the active rTMS intervention.

DETAILED DESCRIPTION:
The primary objectives of this project are as follows:

1. To assess the efficacy TMS in PSD. We hypothesize that there will be a decrease in the HAMD score in patients receiving TMS
2. To assess the feasibility of an accelerated protocol using rTMS in patients with acute to subacute stroke and co-existing PSD. We hypothesize that the accelerated protocol will promote compliance in our patient population and that the administration of this intervention is feasible.
3. To assess the safety of rTMS in patients with acute to subacute stroke. We hypothesize that the side effects of TMS will be minimal and the therapy will be well-tolerated and safe in individuals with recent strokes and co-existing PSD.

ELIGIBILITY:
Inclusion Criteria:

* Between the ages of 22-85 years old
* Radiographic evidence of acute or subacute stroke
* Ischemic stroke diagnosed within the last 2 weeks to 6 months
* HAMD depression score 8 or greater
* Able to provide written informed consent
* Agree to participate in all study procedures

Exclusion Criteria:

* Metallic objects or neurostimulators implanted intracranially
* Stroke in the area of stimulation
* Current thoughts of SI or self-harm as assessed by the M.I.N.I. Suicide Scale score > 8
* ASRM (Altman Self Rating Mania Scale) score > 6 (6 or above indicates likelihood of manic symptoms)
* Current use of illicit substances
* Known history of epilepsy or seizure disorder
* Clinically significant EKG abnormalities including QTC prolongation >450 ms in men or >480 ms in women

Ages: 22 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 6 (Actual)
Dates: Start 2018-10-24 (Actual); Primary Completion 2020-06-30 (Actual); Study Completion 2020-06-30 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- West Virginia University, Morgantown, West Virginia, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Frey J, Najib U, Lilly C, Adcock A. Novel TMS for Stroke and Depression (NoTSAD): Accelerated Repetitive Transcranial Magnetic Stimulation as a Safe and Effective Treatment for Post-stroke Depression. Front Neurol. 2020 Aug 11;11:788. doi: 10.3389/fneur.2020.00788. eCollection 2020. PMID 32849235

RESULTS

PARTICIPANT FLOW:
Groups:
- TMS: NeuroStar TMS Therapy: Open label single arm study to determine safety and effectiveness of TMS for post stroke depression
  TMS: NeuroStar TMS Therapy
Period: Overall Study
Arm/Group | TMS: NeuroStar TMS Therapy
Started | 6
Completed | 6
Not Completed | 0

BASELINE CHARACTERISTICS:
Groups:
- Open Label: Open label single arm study to determine safety and effectiveness of TMS for post stroke depression
  TMS: NeuroStar TMS Therapy
Arm/Group | Open Label
Number analyzed (Participants) | 6
Age, Continuous [Mean (Standard Deviation); unit: years] | 66.33 (4.97)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1
  Male | 5
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Adverse Events
Description: Count of Adverse Events Reported during follow up
Time Frame: After Day 1 of rTMS treatment
Measure: Count of Participants; unit: Participants
Arm/Group | Open Label
Number analyzed (Participants) | 6
Participants | 0

2. Primary Outcome: Number of Participants With Adverse Events
Description: Count of Adverse Events Reported during follow up
Time Frame: After Day 2 of rTMS treatment
Measure: Count of Participants; unit: Participants
Arm/Group | Open Label
Number analyzed (Participants) | 6
Participants | 0

3. Primary Outcome: Number of Participants With Adverse Events
Description: Count of Adverse Events Reported during follow up
Time Frame: After Day 3 of rTMS treatment
Measure: Count of Participants; unit: Participants
Arm/Group | Open Label
Number analyzed (Participants) | 6
Participants | 0

4. Primary Outcome: Number of Participants With Adverse Events
Description: Count of Adverse Events Reported during follow up
Time Frame: After Day 4 of rTMS treatment
Measure: Count of Participants; unit: Participants
Arm/Group | Open Label
Number analyzed (Participants) | 6
Participants | 0

5. Primary Outcome: Number of Participants With Adverse Events
Description: Count of Adverse Events Reported during follow up
Time Frame: 3 months following neurostimulation
Measure: Count of Participants; unit: Participants
Arm/Group | Open Label
Number analyzed (Participants) | 6
Participants | 0

6. Primary Outcome: Number of Participants With Adverse Events
Description: Count of Adverse Events Reported during follow up
Time Frame: 6 months following neurostimulation
Measure: Count of Participants; unit: Participants
Arm/Group | Open Label
Number analyzed (Participants) | 6
Participants | 0

7. Primary Outcome: Number of Participants With Adverse Events
Description: Count of Adverse Events Reported during follow up
Time Frame: 12 months following neurostimulation
Measure: Count of Participants; unit: Participants
Arm/Group | Open Label
Number analyzed (Participants) | 6
Participants | 0

8. Primary Outcome: Depressive Symptoms as Rated by the Hamilton Depression Rating Scale
Description: Depressive symptoms as rated by the Hamilton Depression Rating Scale. Measure of severity of depression -total score of Hamilton Depression Scale ranges from 0 (no depression) to 60 (worst depression possible)
Time Frame: Depressive symptoms will be quantified before the rTMS stimulation protocol
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Open Label
Number analyzed (Participants) | 6
score on a scale | 15.50 (2.81)

9. Primary Outcome: Depressive Symptoms as Rated by the Hamilton Depression Rating Scale
Description: as for outcome 8
Time Frame: Depressive symptoms will be quantified immediately after the 4 days of rTMS stimulation.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Open Label
Number analyzed (Participants) | 6
score on a scale | 4.17 (0.98)

10. Primary Outcome: Depressive Symptoms as Rated by the Hamilton Depression Rating Scale
Description: as for outcome 8
Time Frame: Depressive symptoms will be quantified 3 months after completion of the rTMS stimulation protocol.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Open Label
Number analyzed (Participants) | 6
score on a scale | 3.50 (2.66)

11. Primary Outcome: Depressive Symptoms as Rated by the Hamilton Depression Rating Scale
Description: as for outcome 8
Time Frame: Depressive symptoms will be quantified 6 months after completion of the rTMS stimulation protocol.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Open Label
Number analyzed (Participants) | 6
score on a scale | 5 (3.05)

12. Primary Outcome: Depressive Symptoms as Rated by the Hamilton Depression Rating Scale
Description: as for outcome 8
Time Frame: Depressive symptoms will be quantified 12 months after completion of the rTMS stimulation protocol.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Open Label
Number analyzed (Participants) | 6
score on a scale | 4.667 (5.022)

ADVERSE EVENTS:
Time Frame: 1 year
Description: Adverse events will be monitored via the adverse events screening forms and patients will be routinely asked if they are experiencing any side effects during the treatment process.
Arm/Group | Open Label
All-Cause Mortality (participants affected / at risk) | 0/6
Serious Adverse Events (participants affected / at risk) | 0/6
Other Adverse Events (participants affected / at risk) | 0/6

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol, Statistical Analysis Plan, and Informed Consent Form (2019-09-25): https://cdn.clinicaltrials.gov/large-docs/43/NCT04093843/Prot_SAP_ICF_000.pdf